CLINICAL TRIAL: NCT00424918
Title: Generation-Fit, a Pilot Study of Youth in Maine Middle Schools Using an "Exerlearning" Dance Video Game to Promote Physical Activity During School
Brief Title: "Generation Fit and Exerlearning With In the Groove"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Ann Maloney MD, MMCRI
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MMCRI-3000
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Obesity
Keywords: Dance; Peers; middle school-based; feasibility
MeSH Terms: conditions — Obesity | interventions — Exercise

INTERVENTIONS:
Behavioral: Physical Activity, reduced sedentary behavior

SUMMARY:
In middle schools participating in a statewide program called "Take Time", we are randomizing youth to a 10-12 week intervention using the dance mat games on the Playstation2 (like Dance Dance Revolution). This program is testing feasibility of using the dance mats as a way to increase activity during the school day. We are using "Groove Masters" as a peer-mentored mechanism to keep track of the activity of youth in the intervention compared to the control group. Our main objective is increase in activity time.

DETAILED DESCRIPTION:
We met with administrators and teachers and obtained consent and assent for this study. After assessing baseline measures (end-of-grade test scores, absenteeism, Pediatric Quality of Life, physical fitness, GEMS Activity Rating Scale, Dennison's measure of sedentary screen time, Physical Activity Enjoyment Scale, BMI%ile, (with a small subset assayed for fasting lipids and glucose, with a smaller subset wearing ActiGraphs for objective measures of activity) we randomized to the intervention or control group.

In our intervention, youth play a dance game at school called "In the Groove", with the goal of 40 additional minutes each week of physical activity during the school hours.

We will obtain change scores and compare the groups to find an effect size for future studies, this this proves acceptable and feasible in Maine schools.

ELIGIBILITY:
Inclusion Criteria:

* Take Time middle school in Maine with consent/assent

Exclusion Criteria:

* Any condition that prevents a child from doing physical activity on the dance mat like photic seizures, broken leg, blindness.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Estimated)
Dates: Start 2006-09 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Minutes of activity added in school day.

SECONDARY OUTCOMES:
Quality of Life change scores
Relation to test scores, absenteeism
Fitness change scores
Change in biological endpoints
Others

CONTACTS AND LOCATIONS:
Overall Officials: Ann E Maloney, MD, Principal Investigator — Research Attending
Locations (1):
- Portland, Portland, Maine, United States

REFERENCES:
- [Background] Lanningham-Foster L, Jensen TB, Foster RC, Redmond AB, Walker BA, Heinz D, Levine JA. Energy expenditure of sedentary screen time compared with active screen time for children. Pediatrics. 2006 Dec;118(6):e1831-5. doi: 10.1542/peds.2006-1087. PMID 17142504
- See also: Take Time — http://www.maine-nutrition.org/Projects/MNTT.htm